CLINICAL TRIAL: NCT04724187
Title: Comparison of Intrauterine Misoprostol Plus Intravenous Oxytocin Versus Intravenous Oxytocin Alone for Prevention of Primary Postpartum Haemorrhage in Population of Bhara Kahu.
Brief Title: Prevention of Primary Postpartum Haemorrhage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Islamabad Medical and Dental College (Other)
Responsible Party: Principal Investigator, Afnan Rizwan, Assistant professor, Islamabad Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ARizwan
Record Dates: First submitted 2020-10-28; First posted 2021-01-26 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Primary; Post Partum Hemorrhage
Keywords: primary,oxytocin,; postpartum haemorrhage; mesoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Arthotec; Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrauterine misoprostol and oxytocin (Experimental): there will be added effect of misoprostol to stimulate uterine contraction along with oxytocin
  Interventions: Drug: Misoprostol; Drug: Oxytocin
- oxytocin (Active Comparator): only oxytocin will stimulate uterine contraction
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — it is prostaglandin E1 .
  Other Names: Arthotec
  Arms: intrauterine misoprostol and oxytocin
Drug: Oxytocin — it stimulates uterine contractions
  Other Names: syntocinon

SUMMARY:
Postpartum hemorrhage, is one of the most deadly complication of pregnancy worldwide and major cause of maternal mortality especially in third world countries .1 PPH affects about 5% of all women giving birth around the world 2 .Primary PPH is defined as ≥500 mL blood loss after vaginal delivery or ≥1000 mL after CS delivery within 24 hours after birth1 . Globally, almost one quarter of all maternal deaths are linked with PPH 2. Due to the high prevalence of anemia among pregnant women in low-resource settings, the outcome of PPH is often deteriorated, resulting in damaging health consequences 3. Roughly in 70% of cases of primary pph are due to uterine atony11. Uterine atony is due to loss of contraction and retraction of myometrial muscle fibers can lead to severe hemorrhage and shock. There are several reasons behind uterine atony including maternal anemia, fatigue due to prolong labour and rapid forceful labour. Blood loss is double in caesarean section due to use of increased anesthetic agents4. According to WHO use of oxytocin (10 IU, IM /IV) is recommended for prevention of PPH for all births2. Despite its effectiveness, 10-40% of cases need additional uterotonics to ensure good uterine contraction.5 After oxytocin , Misoprostol is increasingly known as a potential treatment option for PPH 5 .Misoprostol is easily available , rapid acting , and cost effective with minimal side effects, however in caesarean section owing to the effect of anesthesia limits its use . In recent study conducted at Egypt, oxytocin plus misoprostol (study group) is compared with oxytocin alone (control group). Incident of pph was significantly lower in study group (p=0.018), as in study group (1.33%) than control group (6.67%)8. Misoprostol is an autacoid substance and act better if placed closed to target organ 9. Several routes of misoprostol, with or without oxytocin, and its result on intrapartum and postpartum hemorrhage are described in the literature. The practice of misoprostol by the intrauterine route during caesarean section is under trial.10. Aim of study is to observe the effectiveness of intrauterine misoprostol in addition to oxytocin to minimize the blood loss during caesarean section.

DETAILED DESCRIPTION:
Data will be collected from all the patients full filling inclusion criteria on especially designed Performa after informed consent of patient, demographic data will be collected on that preform Patients will be randomized and divide in to two groups group A ( study group ) and group B (controls) , patients under group A will be given 600 microgram misoprostol through intra uterine route during lower segment caesarean section after delivery of placenta in addition to oxytocin 10IU IV and Group B (control) only oxytocin 10IU IV will be given according to WHO protocol .In both groups pre-operative hemoglobin done within 24 hours before the surgery will be recorded and compared with post-operative hemoglobin estimated by blood sample taken 48 hours after the surgery .Mean blood loss during caesarean section will be documented by counting the number of towels , need of additional drugs (repeat oxytocin, tranexamic acid, additional misoprostol) ,time of contractility of uterus, blood transfusion, side effects of misoprostol that is fever, shivering, nausea, vomiting will be recorded 24 hours postoperative period.

All the collected data will be entered and analyzed by SPSS v. 21. Mean and standard deviation will be calculated for quantitative variables like age, gestational age, BMI, pre and post Hb, and blood loss during caesarean section. Frequencies along with percentages will be presented for qualitative variables like need of additional drugs, and side effects of misoprostol (fever, shivering, nausea, vomiting). Paired sample t-test will be used to compare pre and post Hb levels of both groups. Independent sample t-test will be applied to compare post Hb level, blood loss between both groups. Chi-square test will be employed to compare side effects (fever, shivering, nausea, vomiting) between both groups. P-value ≤ 0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria

* 1. All LSCS including emergency and elective 2. Full term pregnancy >37 week

Exclusion Criteria:

* 1. All vaginal deliveries 2. Patients with bleeding or clotting disorders 3. Maternal cardiac, renal, hepatic diseases 4. Morbidly adherent placentas 5. Preterm deliveries

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — reproductive age group 18-40years
Enrollment: 180 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
measurement of haemoglobin level to assess the blood loss | six months
  haemoglobin will be measured preoperatively and postoperatively to minimize the blood loss during cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Islamabad medical and Dental College, Islamabad, Federal, Pakistan